CLINICAL TRIAL: NCT02116907
Title: An Open-Label, Single-Dose Study to Determine the Metabolism and Elimination of 14C-Perampanel in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-A001-049; 2010-018518-56 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Healthy; Male Subjects
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perampanel (Experimental): 14C-labeled perampanel dissolved in ethanol and administered using a capsule formulation in a single dose, one day
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007 — 14C-labeled perampanel dissolved in ethanol and administered using a capsule formulation in a single dose, one day

SUMMARY:
This is an open-label, single-dose study in healthy male subjects. The study will have 2 phases: Pretreatment and Treatment. The Pretreatment Phase will last up to 21 days and will consist of a Screening Period and a Baseline Period, during which each subject's study eligibility will be determined and baseline assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male 18 to 55 years, inclusive, at the time of informed consent
2. Body mass index (BMI) of 18 to 30 kg/m2, inclusive, at Screening
3. Must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must not be of childbearing potential or must be practicing highly effective contraception throughout the study period and for 90 days after study drug discontinuation. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.
4. Provide written informed consent
5. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

1. Participated in a 14C research study within the 6 months before Day-2. The total exposure from this and any previous study must be within the recommended levels considered safe (per 21 Code of Federal Regulations [CFR] 361.1)
2. Exposure to clinically significant radiation within 12 months before Day-2
3. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical attention within 4 weeks of dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of 14C as a cumulative percent of the radiolabeled dose and the identification and quantification of metabolites in humans in vivo after administration of a single dose of radiolabeled 14C-perampanel in healthy male subjects. | Approximately 14 Weeks
  These will be guided by analysis of 14C-perampanel, perampanel, and metabolites in the biological matrices.
Pharmacokinetics of total radioactivity and E2007: Maximum observed concentration (Cmax) | Approximately 14 Weeks
Pharmacokinetics of total radioactivity and E2007: time to reach maximum (peak) concentration following drug administration (tmax) | Approximately 14 Weeks
Pharmacokinetics of total radioactivity and E2007: AUC(0-24h) | Approximately 14 Weeks
  Area under the concentration x time curve from time 0 to 24 hours
Pharmacokinetics of total radioactivity and E2007: AUC(0-t) | Approximately 14 Weeks
  Area under the concentration x time curve from time 0 to time of last measurable concentration
Pharmacokinetics of total radioactivity and E2007: AUC(0-inf) | Approximately 14 Weeks
  Area under the concentration x time curve from time 0 to infinity
Pharmacokinetics of total radioactivity and E2007: terminal elimination half-life (t1/2) | Approximately 14 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States